CLINICAL TRIAL: NCT05635383
Title: Investigation of the Frequency and Causes of Rebound Pain Phenomenon After Peripheral Nerve Blocks
Brief Title: REBOUND PAIN AFTER PERIPHERAL NERVE BLOCKS
Status: Completed | Type: Observational
Sponsor: Diskapi Yildirim Beyazit Education and Research Hospital (Other Government)
Responsible Party: Principal Investigator, Funda Atar, Principal Investigator, Diskapi Yildirim Beyazit Education and Research Hospital
Other Study IDs: 9.5.2022 137/01
Record Dates: First submitted 2022-11-23; First posted 2022-12-02 (Actual); Last update posted 2024-03-28 (Actual); Status verified 2024-03

CONDITIONS: Pain; Block
Keywords: REBOUND PAIN; PERIPHERAL NERVE BLOCKS; analgesia
MeSH Terms: conditions — Pain; Bites and Stings; Agnosia

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: PERIPHERAL NERVE BLOCK — Observation of rebound pain after peripheral nerve block application

SUMMARY:
In recent years, the use of regional anesthesia techniques as part of multimodal analgesia strategies to maximize pain control in patients has reduced opioid requirements and promoted early mobility and rehabilitation in the perioperative period. Regional anesthesia has benefits, mainly peripheral nerve blocks (PNB), muscle relaxation, and postoperative analgesia, thus allowing for control of postoperative pain and early discharge from the hospital. In addition, using PNB techniques provides:

Hemodynamic stability. Reduced need for a post-anesthetic care unit (PACU). Reduced unplanned hospitalization for pain control. Less airway management. Reduced incidence of opioid-related adverse events. Greater patient satisfaction

The main feature of rebound pain is that it is severe pain, within 8-24 hours after PNB. It usually remains severe for 2-6 hours, but the subsequent pain trajectory is consistent with the recovery process expected at surgical intervention. Therefore, rebound pain is temporary and different from persistent post-surgical pain (PPSP).

Rebound pain often occurs at night. However, this is probably related to the 8 to 12-hour duration of most single-injection PNBs and the completion of most elective surgeries during daylight hours.

DETAILED DESCRIPTION:
This study aims to reveal the rebound pain profile, determine the risk factors, and contribute to developing strategies that can prevent rebound pain.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged >18 years who underwent orthopedic surgery with the peripheral nerve block

Exclusion Criteria:

* Patients who did not want to participate in the study
* dementia
* severe psychiatric or cognitive dysfunction
* coagulopathy
* neuropathic disorder
* local anesthetic allergy
* serious heart-lung disease
* chronic opioid use

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients aged >18 years who underwent orthopedic surgery with the peripheral nerve block will be included in the study.
Sampling Method: Probability Sample
Enrollment: 386 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-03-12 (Actual)

PRIMARY OUTCOMES:
incidence of rebound pain | perioperative period
  Rebound pain-defined as transient acute postoperative pain within 12-24hrs that ensues following resolution of sensory blocked.

SECONDARY OUTCOMES:
rebound pain risk factors | perioperative period
  such as age, gender, and presence of preoperative pain.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - University of Medical Science, Yıldırım Beyazıt Training and Research Hospital, Ankara
  - Diskapi Yildirim Beyazit Education and Research Hospital, Ankara

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Williams BA, Bottegal MT, Kentor ML, Irrgang JJ, Williams JP. Rebound pain scores as a function of femoral nerve block duration after anterior cruciate ligament reconstruction: retrospective analysis of a prospective, randomized clinical trial. Reg Anesth Pain Med. 2007 May-Jun;32(3):186-92. doi: 10.1016/j.rapm.2006.10.011. PMID 17543812
- [Background] Gramke HF, de Rijke JM, van Kleef M, Kessels AG, Peters ML, Sommer M, Marcus MA. Predictive factors of postoperative pain after day-case surgery. Clin J Pain. 2009 Jul-Aug;25(6):455-60. doi: 10.1097/AJP.0b013e31819a6e34. PMID 19542791
- [Result] Lavand'homme P. Rebound pain after regional anesthesia in the ambulatory patient. Curr Opin Anaesthesiol. 2018 Dec;31(6):679-684. doi: 10.1097/ACO.0000000000000651. PMID 30124544